CLINICAL TRIAL: NCT02086071
Title: Feasibility of New Biological and Histological Samples at Progression for Patients With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC)
Brief Title: Feasibility of re Biopsies at Progression
Acronym: GFPC-REBIOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GFPC-REBIOP
Record Dates: First submitted 2013-10-06; First posted 2014-03-13 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2014-03

CONDITIONS: Lung Cancer
Keywords: REBIOP re-biopsies advanced or metastatic NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Re biopsies feasibility (Other): the Interest of the study is to evaluate the feasibility of the re biopsy; the re biopsy is done if the patient agrees to perform it.
  Interventions: Procedure: re biopsy

INTERVENTIONS:
Procedure: re biopsy — re biopsy depending on the location of the pathology

SUMMARY:
Feasibility of new biological and histological samples at progression in patients with advanced or metastatic Non Small Cell Lung Cancer (NSCLC).

A recent paper from Professor Sequist and coll. has depicted the resistance mechanisms as Thréonine790Methionine (T890M) mutation oncogene cMet (CMet) amplification. Re-biopsies showed in 14% of cases the transition between NSCLC to Small Cells Lung Cancer (SCLC). In 3 patients, resistance mechanisms have disappeared and they became again sensitive to Tyrosine Kinase Inhibitors (TKIs). It is mandatory to have a better description to natural history of the disease. This study will be conducted by the French Group of Pneumology-Oncology (Groupe Français de Pneumo Cancérologie (GFPC)) up to 100 patients during 18 Months. Each center will have to define if re-biopsies are possible or not and explain why not.

DETAILED DESCRIPTION:
ABSTRACT PROMOTOR GFPC

MAIN INVESTIGATORS Pr Vergnenegre Alain, Dr Dujon Cécile, Pr Rosell Rafael TITLE Feasibility of new biological and histological samples at progression in patients with advanced or metastatic Non Small Cell Lung Cancer (NSCLC)

JUSTIFICATION / BACKGROUND In NSCLC, recent progresses have been reached, with better outcome in terms of survival without relapse, response rate, and improvement of Qualify of Life (QoL). In the detail, patients with mutations of Epidermal Growth Factor Receptor (EGF-R) are sensitive to tyrosine kinase inhibitors (TKIs).

1. Patients with EGF-R mutation Response and disease control are frequently achieved on some long period of time but, in the majority of cases, resistances appear around a period of 12 months after the diagnosis. One of the major resistance mechanisms is the onset of T790M mutation, which induces a non sensitivity to TKIs. At the opposite, some recent papers have depicted that, after a free interval, resistant tumor can be responder in a second phase to TKIs]. The type of the mutation has different consequences on the disease evolution. A recent paper from Pr. Sequist and coll. has depicted the resistance mechanisms as mutation T790M or oncogene cMet (CMet) amplification. Re-biopsies showed in 14% of cases the transition between NSCLC to SCLC. In 3 patients, resistance mechanisms have disappeared and they became again sensitive to TKIs. It is mandatory to have a better description to natural history of the disease.
2. Patients without EGF-R mutation The knowledge of genetic characteristics is currently needed to perform an inclusion in some research protocol.

TRIAL DESIGN Translational study with iterative biopsies.

OUTCOMES CRITERIA Principal outcome Feasibility of re-biopsies

Secondary outcomes

* analyses and types of resistances,
* time until metastasis disappearance
* correlations with disease management
* biological history of the disease.

INCLUSION CRITERIA All the patient more than 18 years old, with advanced or metastatic NSCLC.

NON INCLUSION CRITERIA

* SCLC, neuroendocrine carcinoma,
* Patients with judicial protection or deprived of liberty

PROCEDURES

A paper CRF will be recorded with data on :

* Patients's characteristics,
* Tumor Node Metastasis classification (TNM) and stage,
* Number of metastasis and location at the diagnosis,
* First line treatment: surgery, radiotherapy, chemotherapy,
* Date of EGF-R status response,
* Date of relapse,
* Type of procedures,
* Treatment for second and third line management

NUMBER OF PATIENTS 100 patients NUMBER OF CENTRES 20 centres DURATION 18 months

PRACTICAL ORGANIZATION IN EACH CENTER Each center will have to define if re-biopsies are possible or not (and explain why not). Some localisations are difficult to biopsy like bone metastasis or deep brain metastasis. A bronchial fiberscopy will be systematically performed to search an endoluminal lesion, which could allow 3 to 5 tissue samples. When possible, liver, adrenal gland, superficial brain metastases will be analysed after the relapse.

1. For patients with EGF-R mutation The samples will be prepared with the usual technic of each center. The corresponding slides have to be send to spanish laboratory (Pr R Rosell, Badalona hospital) A comparison between patients with impossible re-biopsies and the final patients group will be performed.
2. For patients without EGF-R mutation the usual practice will be used with biological platforms

BIOLOGICAL PROCEDURES

1. Patients with EGF-R mutation Biological markers analysis will be coordinated by Catalan Institute of Oncology.
2. Patients without EGF-R mutation: usual biological analysis will be performed in the local platform.

STATISTICAL ANALYSES A description of each items will be performed in terms of frequence, range, mean and median. Correlation between biological markers will be assessed by non parametric tests Wilcoxon or Mann-Whitney.

POSSIBLE APPLICATIONS

* a better knowledge of resistance mechanisms in EGF-R mutated patients
* a better knowledge of genetical and molecular history of these diseases
* a better management according to biological changes and evolution

ELIGIBILITY:
Inclusion Criteria:

* All the patient more than 18 years old with advanced or metastatic NSCLC in progression after one or more treatment by chemotherapy.

Exclusion Criteria:

* SCLC, neuroendocrine carcinoma,
* Patients with judicial protection or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of re-biopsies | 18 months / 100 patients
  Feasibility of re-biopsies in patients with advanced or metastatic NSCLC after progression of disease under treatment. If the re-biopsy could not be performed : reason of no re-biopsy. If the biopsy could be performed : site and method of rebiopsy.

SECONDARY OUTCOMES:
Type of resistance | 18 months/100 patients
  Comparison of types and numbers of resistances before treatment (on the first biopsy) and after treatment (on the re-biopsy). Appearance and/or disappearance of some resistances.
Disease management | 18 months / 100 patients
  Description of population: age, performance status, smoking status, sex (number, medium, maximum, minimum). Description of treatment: chemotherapy (type and products), radiotherapy (site), surgery (site)
Biological history of the disease | 18 months / 100 patients
  Description and comparison of histology on the first biopsy and on the rebiopsy

CONTACTS AND LOCATIONS:
Overall Officials: DUJON Cécile, MD, Principal Investigator — CENTRE HOSPITALIER André MIGNOT VERSAILLES FRANCE
Locations (9):
- France (9):
  - Centre Hospitalier Universitaire, Angers
  - Centre Hospitalier du Morvan, Brest
  - Centre François Baclesse, Caen
  - Site 04, Gap
  - Hospital du Cluzeau, Limoges
  - Site 25, Mantes-la-Jolie
  - Site 06, Marseille
  - Hospital Saint Antoine, Paris
  - Site 20, Rennes